CLINICAL TRIAL: NCT00782418
Title: A Randomized Clinical Trial to Study Glucose Dependent Insulin Secretion Methodologies in Healthy Lean Male Subjects
Brief Title: A Study to Compare Methodologies for Assessing Glucose-Dependent Insulin Secretion (0000-104)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-104; 2008_568
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2010-04-06 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-11

CONDITIONS: The Methodology Assessment of Glucose Dependent Insulin Secretion
MeSH Terms: interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): exenatide 5mcg
  Interventions: Drug: Comparator: exenatide
- 2 (Active Comparator): exenatide 1.5mcg
  Interventions: Drug: Comparator: exenatide
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: exenatide — exenatide in two 5mcg subcutaneous doses 120 minutes apart, followed by either HGC or GGI. After a 14 day washout period two additional 5mcg doses will be administered, followed by HCG or GGI.
  Other Names: Byetta
  Arms: 1
Drug: Comparator: exenatide — exenatide in two 1.5mcg subcutaneous doses 120 minutes apart, followed by either HGC or GGI. After a 14 day washout period two additional 1.5mcg doses will be administered, followed by HCG or GGI.
  Other Names: Byetta
  Arms: 2
Drug: Comparator: Placebo — 5% osmitrol in two 60 mcL subcutaneous doses 120 minutes apart, followed by either HGC or GGI. After a 14 day washout period two additional 60 mcL doses will be administered, followed by HCG or GGI.
  Arms: 3

SUMMARY:
This study will compare graded glucose infusion (GGI) to the hyperglycemic clamp (HGC) for assessment of glucose-dependent insulin secretion (GDIS) using exenatide as a probe.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Body Mass Index (BMI) of less than or equal to 26 kg/m2 at screening
* Subject is judged to be in good health
* Subject has been a nonsmoker for at least 3 months
* Subject is willing to avoid strenuous physical activity for the duration of the study

Exclusion Criteria:

* Subject has a history of high blood pressure requiring treatment
* Subject has a history of diabetes or a family history of diabetes mellitus
* Subject is unable to discontinue all prescription and non-prescription drugs for duration of study
* Subject consumes more than 3 alcoholic beverages per day
* Subject consumes more than 6 servings of caffeinated beverages per day (1 serving = 120mg caffeine)
* Subject has had major surgery or has donated or loss 1 unit of blood within 4 weeks of screening
* Subject has multiple and/or severe allergies to foods or drugs
* Subject is a regular user of illegal drugs
* Subject is unwilling or unable to consume the standardized meals during the study and/or is on a carbohydrate restricted diet

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shankar SS, Shankar RR, Mixson LA, Miller DL, Chung C, Cilissen C, Beals CR, Stoch SA, Steinberg HO, Kelley DE. Linearity of beta-cell response across the metabolic spectrum and to pharmacology: insights from a graded glucose infusion-based investigation series. Am J Physiol Endocrinol Metab. 2016 Jun 1;310(11):E865-73. doi: 10.1152/ajpendo.00527.2015. Epub 2016 Apr 12. PMID 27072496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered: 19-Sep-2008
  Last Patient, Last Visit: 05-Mar-2009
  1 site
Pre-assignment Details: Inclusion criteria: Subjects with a Body Mass Index (BMI) of ≤26 kg/m2
  Exclusion criteria: History of diabetes or family history of diabetes.
  Subjects on a carbohydrate restricted diet.
  An amendment added 8 subjects to go before study completion and instituted down dosing for subjects assigned to exenatide 5 μg in the HGC period to placebo
Groups:
- HGC - Exenatide 5 μg: Hyperglycemic Clamp (HGC): Treatment Group Exenatide 5 μg
- HGC - Exenatide 1.5 μg: Hyperglycemic Clamp: Treatment Group Exenatide 1.5 μg
- HGC - Placebo: Hyperglycemic Clamp: Treatment Group Placebo
- Exenatide 5 ug Down Dosed to Placebo (HGC): Hyperglycemic Clamp: Treatment Group Exenatide 5 ug down dosed to placebo
- GGI - Exenatide 5 μg: Graded Glucose Infusion (GGI): Treatment Group Exenatide 5 μg
- GGI - Exenatide 1.5 μg: Graded Glucose Infusion: Treatment Group Exenatide 1.5 μg
- Placebo (HGC or GGI): Hyperglycemic Clamp or Graded Glucose Infusion: Treatment Group Placebo
Period: Period 1 Procedure/Treatment Groups
Arm/Group | HGC - Exenatide 5 μg | HGC - Exenatide 1.5 μg | HGC - Placebo | Exenatide 5 ug Down Dosed to Placebo (HGC) | GGI - Exenatide 5 μg | GGI - Exenatide 1.5 μg | Placebo (HGC or GGI)
Started | 3 | 4 | 4 | 2 | 5 | 5 | 4
Completed | 1 | 4 | 4 | 2 | 4 | 4 | 4
Not Completed | 2 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study placed on temporary hold | 1 | 0 | 0 | 0 | 1 | 1 | 0
Period: Period 2 Procedure/Treatment Groups
Arm/Group | HGC - Exenatide 5 μg | HGC - Exenatide 1.5 μg | HGC - Placebo | Exenatide 5 ug Down Dosed to Placebo (HGC) | GGI - Exenatide 5 μg | GGI - Exenatide 1.5 μg | Placebo (HGC or GGI)
Started | 3 | 4 | 4 | 1 | 3 | 4 | 4
Completed | 3 | 4 | 4 | 1 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients from all arms
Arm/Group | All Patients
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (9.1)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.3 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Secretion Rate (ISR) Normalized to Ambient Plasma Glucose
Description: Comparison of Glucose Dependent Insulin Secretion (GDIS) measured after HGC at steady-state to GDIS measured after GGI at the highest glucose infusion rate.
  Insulin Secretion Rate (ISR)/ Blood Glucose (BG)
Time Frame: Steady-state of HGC: 90 - 120 minutes post dose; highest glucose infusion rate of GGI: 120 - 160 minutes post dose
Population: All subjects treated
Measure: Geometric Mean (Full Range); unit: (ng/min) / (mg/dL)
Groups:
- GGI - Placebo: Graded Glucose Infusion: Treatment Group Placebo
Arm/Group | HGC - Exenatide 5 μg | HGC - Exenatide 1.5 μg | HGC - Placebo | GGI - Exenatide 5 μg | GGI - Exenatide 1.5 μg | GGI - Placebo
Number analyzed (Participants) | 6 | 8 | 11 | 6 | 9 | 8
(ng/min) / (mg/dL) | 2.14 [1.52 to 2.52] | 1.49 [0.78 to 2.16] | 0.53 [0.19 to 0.73] | 2.95 [0.94 to 3.88] | 2.07 [0.82 to 3.30] | 0.71 [0.10 to 1.22]
Statistical Analysis 1: Comparison: HGC - Exenatide 5 μg vs HGC - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided, alpha=0.05; Least Squares Mean = 1.60, 90% CI [1.29 to 1.92]
Statistical Analysis 2: Comparison: HGC - Exenatide 1.5 μg vs HGC - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; 1-sided, alpha=0.05; Least Squares Mean = 0.95, 90% CI [0.66 to 1.24]
Statistical Analysis 3: Comparison: GGI - Exenatide 5 μg vs GGI - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; 1-sided, alpha=0.05; Least Squares Mean = 2.32, 90% CI [1.57 to 3.06]
Statistical Analysis 4: Comparison: GGI - Exenatide 1.5 μg vs GGI - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; 1-sided, alpha = 0.05; Least Squares Mean = 1.38, 90% CI [0.64 to 2.12]

2. Primary Outcome: Change From Baseline in C-peptide Concentration
Time Frame: Pre and Post glucose infusion
Population: All subjects treated
Measure: Least Squares Mean (Full Range); unit: ng/mL
Arm/Group | HGC - Exenatide 5 μg | HGC - Exenatide 1.5 μg | HGC - Placebo
Number analyzed (Participants) | 6 | 8 | 11
ng/mL | 29.3 [25.2 to 35.1] | 22.6 [14.0 to 34.1] | 6.24 [2.3 to 8.9]
Statistical Analysis 1: Comparison: HGC - Exenatide 5 μg vs HGC - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; 1-side, alpha = 0.05; Least Squares Mean = 23.1, 90% CI [19.2 to 27.0]
Statistical Analysis 2: Comparison: HGC - Exenatide 1.5 μg vs HGC - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; 1-side, alpha = 0.05; Least Squares Mean = 16.4, 90% CI [12.6 to 20.1]

3. Primary Outcome: Change From Baseline in Insulin Concentration
Time Frame: Pre and Post glucose infusion
Population: All subjects treated
Measure: Least Squares Mean (Full Range); unit: μIU(insulin)/mL
Arm/Group | HGC - Exenatide 5 μg | HGC - Exenatide 1.5 μg | HGC - Placebo
Number analyzed (Participants) | 6 | 8 | 11
μIU(insulin)/mL | 592 [445 to 695] | 293 [128 to 597] | 46.5 [16.2 to 123]
Statistical Analysis 1: Comparison: HGC - Exenatide 5 μg vs HGC - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; 1-side, alpha = 0.05; Least Squares Mean = 545.0, 90% CI [451.4 to 638.7]
Statistical Analysis 2: Comparison: HGC - Exenatide 1.5 μg vs HGC - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; 1-side, alpha = 0.05; Least Squares Mean = 246.6, 90% CI [160.9 to 323.3]

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected from the time the consent is signed through the 14 day follow up period after all treatment periods were completed.
Description: AE s were assessed by clinical evaluation including vital signs, physical examination, medical history, clinical laboratory safety assessment (hematology, chemistry, urinalysis), and ECG at timepoints specified in the study. Subjects were queried at each visit for any adverse experiences since the previous visit.
Arm/Group | HGC - Exenatide 5 μg | HGC - Exenatide 1.5 μg | HGC - Placebo | GGI - Exenatide 5 μg | GGI - Exenatide 1.5 μg | GGI - Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 1/7 | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 4/9 | 4/9 | 4/10 | 6/7 | 3/8 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HGC - Exenatide 5 μg (N=9) | HGC - Exenatide 1.5 μg (N=9) | HGC - Placebo (N=10) | GGI - Exenatide 5 μg (N=7) | GGI - Exenatide 1.5 μg (N=8) | GGI - Placebo (N=11)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HGC - Exenatide 5 μg (N=9) | HGC - Exenatide 1.5 μg (N=9) | HGC - Placebo (N=10) | GGI - Exenatide 5 μg (N=7) | GGI - Exenatide 1.5 μg (N=8) | GGI - Placebo (N=11)
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 2 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 5 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood Phosphorus Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disturbance In Attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 0 | 3 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 1
Thrombophlebitis Superficial (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.